CLINICAL TRIAL: NCT02675036
Title: Interceptive Study of Ectopic Eruption of Permanent Maxillary Canine Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Tromso (Other)
Collaborators: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/623/REK
Record Dates: First submitted 2016-01-28; First posted 2016-02-05 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Tooth Eruption,Ectopic
Keywords: ectopiccanine teeth, impacted teeth, tooth eruption, orthodontics
MeSH Terms: conditions — Tooth Eruption, Ectopic; Tooth, Impacted; Exanthema | interventions — Tooth Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary canine tooth (Experimental): Extraction of primary canine tooth
  Interventions: Procedure: Tooth extraction
- Primary canine and primary molar teeth (Experimental): Extraction of primary canine and primary first molar teeth
  Interventions: Procedure: Tooth extraction

INTERVENTIONS:
Procedure: Tooth extraction

SUMMARY:
The purpose of this study is to see whether extraction of the primary canine tooth or extraction of both the primary canine - and the primary first molar tooth is most effective in the treatment of palatally ectopic canine teeth in the maxilla. In addition the study will also measure pain and discomfort in relation to these two treatment alternatives.

DETAILED DESCRIPTION:
Study objectives:

1. Evaluate the effectiveness of concomitant extraction of the maxillary deciduous canine and maxillary deciduous first molar as compared to extraction of the deciduous maxillary canine only as an interceptive measure for improving the eruption path of ectopic maxillary canines.
2. Evaluate whether there is a difference in the use of analgesics, pain and discomfort between the two treatment groups in 1.

Procedure:

After informed consent patients will randomly be assigned to one of two groups. Group1: Extraction of the deciduous canine only Group 2: Extraction of both the deciduous canine and the deciduous first molar

Randomization The block randomization method will be used. Block sizes will randomly vary from 2, 4, 6 and 8. Blocks will be generated from free software at http://www.randomization.com . Allocation concealment is done by enclosing assignments into sequentially numbered envelopes. Envelopes that will have to be torn to open will be used. The randomization process will be done by a staff member at TkNN that is not involved in the trial.

Prior to extractions topical anesthetics will be given for two minutes, before the buccal and palatal infiltration of local anesthetic (1,8 ml dose, 20mg/ml lidocain with 12,5 g/ml epinephrine).

Patients and parents will be given oral postoperative information, including a recommendation to use non-prescription analgesics at their own discretion.

Clinical and Radiographic controls and evaluation:

Patients will be controlled clinically and radiographically (DPT) after 6 and 12 months. If improvement is not detectable after 12 months, alternative treatment will be suggested (surgical exposure, fixed orthodontic appliances, extractions). All cases which do not need alternative approaches will be followed until the tooth is erupted in the mouth.

Sector, alpha angle and d-distance will be measured on DPT-images

Dental anxiety Before any extractions are performed each patient will answer the modified dental anxiety scale (MDAS).

Pain and discomfort When the patients have performed their extractions they will receive two questionnaires, regarding pain and discomfort and use of analgesics, to fulfill at home and return by mail. The first part shall be answered the first evening as the extraction was performed and the second part should be answered one week post extraction.

ELIGIBILITY:
Inclusion Criteria:

* mixed dentition with both primary maxillary canine and primary maxillary first molars present
* palatally ectopic canines present. (palatally ectopic canines will be diagnosed via measurements developed by Ericson and Kurol using DPT images. A canine with and alpha angle of ≥ 25 degrees in sectors 2 through 5, and palatal position observed on intraoral radiographs

Exclusion Criteria:

* previous orthodontic treatment
* any disease not allowing local anesthesia or extraction
* craniofacial syndromes, cleft lip palate
* odontomas, cysts

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change in permant canine tooth position measured by Sector and Alpha angle | 12 months
  Change in Sector and Alpha angle measured on panoramic radiographs will be reported

SECONDARY OUTCOMES:
Pain and discomfort after tooth extraction reported by questionnaire | 1 week after tooth extraction
  Patients pain and discomfort will be reported by VAS - scale

OTHER OUTCOMES:
Full eruption of permanent ectopic canine tooth in to the oral cavity | 12-30 months after primary canine tooth extraction
  The ratio of fully erupted teeth in the oral cavity will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Kerosuo, PhD, Principal Investigator — University of Tromso
Locations (1):
- Tannhelsetjenestens kompetansesenter for Nord-Norge, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benson PE, Atwal A, Bazargani F, Parkin N, Thind B. Interventions for promoting the eruption of palatally displaced permanent canine teeth, without the need for surgical exposure, in children aged 9 to 14 years. Cochrane Database Syst Rev. 2021 Dec 30;12(12):CD012851. doi: 10.1002/14651858.CD012851.pub2. PMID 34967448
- [Derived] Hadler-Olsen S, Sjogren A, Steinnes J, Dubland M, Bolstad NL, Pirttiniemi P, Kerosuo H, Lahdesmaki R. Double vs single primary tooth extraction in interceptive treatment of palatally displaced canines. Angle Orthod. 2020 Nov 1;90(6):751-757. doi: 10.2319/031920-196.1. PMID 33378508